CLINICAL TRIAL: NCT07020819
Title: An Open-Label Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Efficacy, and Safety of a Single Dose of Tanruprubart (Also Commonly Known as ANX005) in Participants With Guillain-Barré Syndrome (GBS) (FORWARD Study)
Brief Title: An Open Label Clinical Study to Evaluate Tanruprubart (Also Commonly Known as ANX005) in Participants With Guillain-Barré Syndrome (FORWARD Study)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Annexon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANX005-GBS-05; 2025-522664-32-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-06; First posted 2025-06-13 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Guillain-Barre Syndrome
Keywords: Guillain-Barre Syndrome; GBS; ANX005; Tanruprubart; FORWARD study
MeSH Terms: conditions — Guillain-Barre Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tanruprubart (Experimental): Participants will receive a single 30 mg/kg intravenous (IV) infusion of tanruprubart on Day 1.
  Interventions: Drug: Tanruprubart

INTERVENTIONS:
Drug: Tanruprubart — Solution for IV infusion.
  Other Names: ANX005

SUMMARY:
The goal of this open label study is to measure pharmacokinetics, pharmacodynamics, early efficacy, and safety of tanruprubart in adult and pediatric participants, in the United States, Canada, and Europe.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of GBS according to the National Institute of Neurological Disorders and Stroke Diagnostic Criteria for GBS.
* Onset of GBS-related weakness ≤10 days before start of infusion on Day 1
* GBS-disability score (DS) score of 3, 4, or 5 at screening and before start of infusion on Day 1.

Key Exclusion Criteria:

* Previous or intended treatment with either plasma exchange or IV immunoglobulin for GBS.
* Diagnosis of a variant of GBS, including Miller Fisher syndrome, Bickerstaff's encephalitis, and overlap syndromes.

Other protocol-defined criteria may apply.

Ages: 12 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Area Under the Tanruprubart Serum Concentration-time Curve to the Last Sample (AUC0-t) | Up to Day 15
Observed Time to Maximum Observed Serum Concentration (Cmax) (Tmax) of Tanruprubart | Up to Day 15

SECONDARY OUTCOMES:
Change From Baseline in Free Component of Complement Complex (C1q) Protein Concentration in Serum | Baseline up to Day 15
Change from Baseline in Medical Research Council (MRC) Sumscore at Week 1 | Baseline, Week 1

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Annexon, Inc.
Locations (4):
- United States (4):
  - Children's Hospital of Orange County, Orange, California
  - University of California Irvine, Orange, California
  - Henry Ford Health, Detroit, Michigan
  - Mayo Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://theforwardstudy.com/